CLINICAL TRIAL: NCT04420351
Title: A Phase ⅢB, Prospective, Randomized, Open Label, Blinded-endpoint, Multicenter Trial of the Efficacy and Safety of Urokinase Thrombolysis Comparing With Antiplatelet Agents for Patients With Minor Stroke.
Brief Title: Thrombolysis of Urokinase for Minor Stroke
Acronym: TRUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Shanghai 10th People's Hospital (Other); General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Bo Song, Chief of neurology department, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017YFC1308202
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Minor Stroke
Keywords: Thrombolysis; Urokinase; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urokinase thrombolysis (Experimental): The patients of intervention group will receive 1 millions units urokinase dissolved by 100 saline through intravenous infusion within 30 minutes.
  Interventions: Drug: Urokinase thrombolysis
- Antiplatelet treatment (Other): The control group will receive antiplatelet agents as decided by the physicians according to Chinese guideline for diagnosis and treatment of acute ischemic stroke 2018
  Interventions: Drug: Aspirin;Clopidogrel

INTERVENTIONS:
Drug: Urokinase thrombolysis — The patients of intervention group will receive 1 millions units urokinase dissolved by 100 saline through intravenous infusion within 30 minutes.
  Other Names: Urokinase
  Arms: Urokinase thrombolysis
Drug: Aspirin;Clopidogrel — The control group will receive antiplatelet agents as decided by the physicians according to Chinese guideline for diagnosis and treatment of acute ischemic stroke 2018.
  Other Names: Antiplatelet treatment
  Arms: Antiplatelet treatment

SUMMARY:
This trial will enroll patients that have been diagnosed with minor stroke, which has occurred within the past 6 hours. TRUST is a prospective multicenter, randomized, blinded-endpoint study to evaluate the efficacy and safety of Urokinase Thrombolysis for patients with minor stroke.

DETAILED DESCRIPTION:
China is currently faced with the heaviest stroke burden due to the tremendous population and susceptibility to cerebrovascular disease. As has been assessed, deaths caused by cerebrovascular disease are three times of cardiovascular disease. Within whole population with cerebrovascular disease, minor stoke have taken a significant part of the disease burden. Thus the population with minor stoke is one of the most important parts in efficient prevention of cerebrovascular disease. According to phase I and II data from national stoke registration in China, 35.25% to 42.23% cases were minor ischemic strokes. However, in clinical practice, the minor ischemic stroke patients are likely to be ignored and some might have poor prognosis. As has been demonstrated by a number of studies, up to one third of the acute non-disabling ischemic stroke without in-time thrombolysis may suffer from disabling or death at 90-day follow-up.

Several studies have demonstrated the potential benefits of thrombolysis compared usually with placebo, including the Third International Stroke Trail ( IST-3, rt-PA to placebo, patients within 3 hours after attack, with blood pressure lower than 185/110mmHg and NIHSS≤5)，National Institute of Neurological Disorders and Stroke rt-PA Stroke Study（ NINDS, rt-PA to placebo, patients with mild ischemic stroke recognized by 5 different definitions）.

Urokinase is a kind of non-selective plasminogen activator, urokinase acted as effective catalyzer in the transferring of both free and protein-binding plasminogen to plasmin, thus inducing thrombolysis. As one of the widely used medication for intravenous thrombolysis in China, urokinase has been suggested the the efficacy and safety for ischemic stroke. With easier availability and lower price, urokinase has provided a promising alternation to patients who need thrombolysis in China, especially in less developed areas. The Chinese guideline for diagnosis and treatment of acute ischemic stroke 2018 has recommended urokinase as an alternation in the treatment of acute ischemic stroke within 6-hour time window as well, if rt-PA is not available or affordable. However, randomized and multicenter clinical trial of urokinase thrombolysis for minor stroke is still vacant, which couldn't provide more persuasive evidence.

TRUST is a prospective multicenter, randomized, single-blind evaluation study to evaluate the efficacy and safety of Urokinase Thrombolysis for patients with minor stroke. The trail will enroll a total of 1002 minor stroke patients within a 6 hour time window with a NIHSS score ≤5 at the time of randomization. Randomization will be 1:1 to Urokinase Thrombolysis (experimental) or Antiplatelet agents (control). Patients will receive 1 million units urokinase dissolved by 100ml saline through intravenous infusion within 30min or oral antiplatelet agents. All patients will undergo CT or MRI before treatment and will undergo the second CT within 36 hours after treatment. Patients will be followed up at 36h, 7d and 90 days. The primary outcome measures including the proportion of patients with a modified Rankin Scale(mRS) of 0 or 1 at 90-day follow-up and the patients with symptomatic intracranial hemorrhage within 36 hours. Secondary outcome measures cover new vascular events, the Progress of MRS score, Neurological impairment, Daily function evaluations, Quality of life assessments, Overall mortality and Adverse events and severe adverse events within 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients: 18-80 years old
2. The time from last seen well to treatment < 6 hours
3. Minor stroke defined as a baseline NIHSS ≤5 at the time of randomization..
4. First onset or pre-stroke mRS≤1
5. Informed consent signed

Exclusion Criteria:

1.Hyperdensity on CT suggesting intracranial hemorrhage

2.Large acute stroke >1/3 middle cerebral artery (MCA) territory visible on CT or MRI

3.Other contraindications of intravenous thrombolysis, including but not limited to:

1. Intracranial tumor, arteriovenous malformation
2. Coma or confirmed as severe stroke by clinical assessment (e.g. NIHSS ≥25) or proper imaging methods
3. With seizure
4. Stroke attack within past three months
5. Heparin administration within 48h before onset, with APTT longer than upper limit
6. Stroke history with diabetes
7. Platelet count ≤100×10^9/L
8. Difficult to control hypertension, defined by systolic pressure ≥185mmHg or diastolic pressure ≥110 mmHg in 3 tests with at least ten minutes interval, under well guided medications.
9. Blood glucose <50mg/dl（2.7mmol/l）or >400mg/dl（22.2mmol/l）
10. Obvious hemorrhage within past 6 months
11. Oral anti-coagulation drug administration (e.g. warfarin) with INR>1.5
12. Intracranial hemorrhage or suspected intracranial hemorrhage (including subarachnoid hemorrhage)
13. Pregnancy or lactation.
14. History of severe CNS damage (e.g. tumor, arterial aneurysm or CNS surgery)
15. Hemorrhagic retinopathy, e.g. diabetes (hemorrhages suggested by optic impairment) or other hemorrhagic ocular lesions.
16. Bacterial endocarditis or pericarditis.
17. Prolonged or traumatic CPR (>2min), puncture in nonstress vessels within past 10 days, such as subclavian vein puncture.
18. Acute pancreatitis.
19. Confirmed ulcerative gastric or intestinal problems within 3 months.
20. Arterial aneurysm or arteriovenous malformation.
21. Any tumor that increase risk of hemorrhage.
22. Severe hepatic diseases, like hepatic failure, liver cirrhosis, portal hypertension, esophageal varices or active hepatitis.
23. Major surgery, severe trauma or craniocerebral trauma within past 10 days.
24. Allergy to any components of urokinase.

4.Severe, fatal diseases with less than 3 month expected survival.

5.Intended to receive standard rt-PA thrombolysis or intravascular therapy.

6.Already participating in other studies that conflict to this study.

7.Unable to accomplish the follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a modified Rankin Scale(mRS) of 0 or 1 at 90-day follow-up | 90 Days
  mRS has 0-6 points, the higher the worse outcome.
Proportion of patients with symptomatic intracranial hemorrhage within 36 hours | 36 hours
  Symptomatic intracranial haemorrhage within 36 hours

SECONDARY OUTCOMES:
Proportion of patients with new vascular events | 90 days
  Proportion of patients with new vascular events within 90 days(Ischemic stroke / hemorrhagic stroke / TIA / myocardial infarction / vascular death)
MRS score | 90 days
  To evaluate the progress of MRS score
The ratio of patients with MRS 0-1 during the last visit in two groups | 90 days
  mRS has 0-6 points, the higher the worse outcome.
Changes in National Institutes of Health Stroke Scale(NIHSS) score | 90 days
  Neurological impairment in two groups (changes in NIHSS score at 90-day follow-up). NIHSS has 0-42 points, the higher the worse outcome.
Barthel index (BI) score | 90 days
  Daily function evaluations(BI score at 90 days). BI has 0-100 points,the higher the bettter outcome.
Quality of life assessments | 90 days
  EuroQol five dimensional questionnaire (EQ-5D scale).
Overall mortality | 90 days
  Overall mortality within 90 days
Adverse events and severe adverse events | 90 days
  Adverse events and severe adverse events in two groups during 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bo Song, MD;PhD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu M, Wu B, Wang WZ, Lee LM, Zhang SH, Kong LZ. Stroke in China: epidemiology, prevention, and management strategies. Lancet Neurol. 2007 May;6(5):456-64. doi: 10.1016/S1474-4422(07)70004-2. PMID 17434100
- [Background] Wu Z, Yao C, Zhao D, Wu G, Wang W, Liu J, Zeng Z, Wu Y. Sino-MONICA project: a collaborative study on trends and determinants in cardiovascular diseases in China, Part i: morbidity and mortality monitoring. Circulation. 2001 Jan 23;103(3):462-8. doi: 10.1161/01.cir.103.3.462. PMID 11157701
- [Background] Liu L, Wang D, Wong KS, Wang Y. Stroke and stroke care in China: huge burden, significant workload, and a national priority. Stroke. 2011 Dec;42(12):3651-4. doi: 10.1161/STROKEAHA.111.635755. Epub 2011 Nov 3. PMID 22052510
- [Background] Smith EE, Fonarow GC, Reeves MJ, Cox M, Olson DM, Hernandez AF, Schwamm LH. Outcomes in mild or rapidly improving stroke not treated with intravenous recombinant tissue-type plasminogen activator: findings from Get With The Guidelines-Stroke. Stroke. 2011 Nov;42(11):3110-5. doi: 10.1161/STROKEAHA.111.613208. Epub 2011 Sep 8. PMID 21903949
- [Background] Barber PA, Zhang J, Demchuk AM, Hill MD, Buchan AM. Why are stroke patients excluded from TPA therapy? An analysis of patient eligibility. Neurology. 2001 Apr 24;56(8):1015-20. doi: 10.1212/wnl.56.8.1015. PMID 11320171
- [Background] Nedeltchev K, Schwegler B, Haefeli T, Brekenfeld C, Gralla J, Fischer U, Arnold M, Remonda L, Schroth G, Mattle HP. Outcome of stroke with mild or rapidly improving symptoms. Stroke. 2007 Sep;38(9):2531-5. doi: 10.1161/STROKEAHA.107.482554. Epub 2007 Aug 2. PMID 17673713
- [Background] Smith EE, Abdullah AR, Petkovska I, Rosenthal E, Koroshetz WJ, Schwamm LH. Poor outcomes in patients who do not receive intravenous tissue plasminogen activator because of mild or improving ischemic stroke. Stroke. 2005 Nov;36(11):2497-9. doi: 10.1161/01.STR.0000185798.78817.f3. Epub 2005 Oct 6. PMID 16210552
- [Background] Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, Subramaniam S, Goyal M, Patil S, Menon BK, Barber PA, Dowlatshahi D, Field T, Asdaghi N, Camden MC, Hill MD; TEMPO-1 Investigators. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015 Mar;46(3):769-74. doi: 10.1161/STROKEAHA.114.008504. Epub 2015 Feb 12. PMID 25677596
- [Background] Khatri P, Tayama D, Cohen G, Lindley RI, Wardlaw JM, Yeatts SD, Broderick JP, Sandercock P; PRISMS and IST-3 Collaborative Groups. Effect of Intravenous Recombinant Tissue-Type Plasminogen Activator in Patients With Mild Stroke in the Third International Stroke Trial-3: Post Hoc Analysis. Stroke. 2015 Aug;46(8):2325-7. doi: 10.1161/STROKEAHA.115.009951. Epub 2015 Jun 23. PMID 26106113
- [Background] National Institute of Neurological Disorders Stroke rt-PA Stroke Study Group. Recombinant tissue plasminogen activator for minor strokes: the National Institute of Neurological Disorders and Stroke rt-PA Stroke Study experience. Ann Emerg Med. 2005 Sep;46(3):243-52. doi: 10.1016/j.annemergmed.2005.02.013. PMID 16126134
- [Background] Khatri P, Kleindorfer DO, Yeatts SD, Saver JL, Levine SR, Lyden PD, Moomaw CJ, Palesch YY, Jauch EC, Broderick JP. Strokes with minor symptoms: an exploratory analysis of the National Institute of Neurological Disorders and Stroke recombinant tissue plasminogen activator trials. Stroke. 2010 Nov;41(11):2581-6. doi: 10.1161/STROKEAHA.110.593632. Epub 2010 Sep 2. PMID 20814000
- [Derived] Tao Y, Gao Y, Zhao L, Xu Y, Jiang C, Liu K, Fang H, Pei L, Wang X, Zhang R, Wu J, Yang J, Han X, Guo H, Xue B, Li J, Liu Y, Gu H, Du K, Cheng X, Dong Q, Wang D, Buonanno FS, Ning M, Xu Y, Song B; TRUST Trial Investigators. Effect of intravenous urokinase vs best medicine treatment on functional outcome for patients with acute minor stroke (TRUST): a randomized controlled trial. BMC Med. 2025 Jan 6;23(1):6. doi: 10.1186/s12916-024-03820-2. PMID 39757192